CLINICAL TRIAL: NCT03666351
Title: A Prospective, Multicentre, Randomized, Open Label, Evaluator-Blind, Phase IV Study to Evaluate the Effect on Improvement of Left Ventricular Hypertrophy by the Control of Blood Pressure in Hypertension Patients With Aortic Valve Disease
Brief Title: Study to Evaluate the Effect on Improvement of LVH by the Control of BP in Hypertension Patients With AV Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM_AMO_401
Record Dates: First submitted 2018-08-20; First posted 2018-09-11 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Aortic Stenosis; Aortic Regurgitation; Hypertension; LVM; Left Ventricular Hypertrophy
Keywords: Aortic Stenosis; Aortic Regurgitation; Hypertension; LVM; Left Ventricular Hypertrophy
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Hypertension; Hypertrophy, Left Ventricular | interventions — Amlodipine; Losartan; amlodipine-losartan drug combination; Tablets

STUDY DESIGN:
Intervention Model Description: A prospective, multicentre, randomized, open label, evaluator-blind study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intensive care group (Experimental): The intensive care group is targeted at ≤ 130 mmHg of systolic blood pressure, and treatment is done by changing the current treatment to the investigational product.
  In case of treatment with the investigational product (IP), the IP titration period is total six months. According to an IP titration scheme(Amlodipine 5 mg or Losartan 50 mg -> Losartan and Amlodipine 5/50 mg -> Losartan and Amlodipine 5/100 mg -> Amlodipine/Losartan/Chlorthalidone 5/100/12.5 mg), IP is successively modified until the target blood pressure is reached, and IP will remain the same after the target blood pressure scope for each group is reached. An IP titration interval is decided by the investigator depending on the subject's condition.
  Interventions: Drug: Amlodipine 5mg; Drug: Losartan; Drug: Losartan and Amlodipine; Drug: Amlodipine/Losartan/Chlorthalidone
- The usual care group (Experimental): The usual care group is targeted at ≤ 140 mmHg of systolic blood pressure, and treatment is done by maintaining the current treatment, adding the investigational product, or changing the current treatment to the investigational product.
  In case of treatment with the investigational product (IP), the IP titration period is total six months. According to an IP titration scheme(Amlodipine 5 mg or Losartan 50 mg -> Losartan and Amlodipine 5/50 mg -> Losartan and Amlodipine 5/100 mg -> Amlodipine/Losartan/Chlorthalidone 5/100/12.5 mg), IP is successively modified until the target blood pressure is reached, and IP will remain the same after the target blood pressure scope for each group is reached. An IP titration interval is decided by the investigator depending on the subject's condition.
  Interventions: Drug: Amlodipine 5mg; Drug: Losartan; Drug: Losartan and Amlodipine; Drug: Amlodipine/Losartan/Chlorthalidone; Drug: current treatment

INTERVENTIONS:
Drug: Amlodipine 5mg — Amlodipine 5 mg
  Other Names: Amodipin Tab.
Drug: Losartan — Losartan Potassium 50 mg
  Other Names: Osartan Tab. 50 mg
Drug: Losartan and Amlodipine — Amlodipine 5 mg/Losartan Potassium 50 mg, Amlodipine 5 mg/Losartan Potassium 100 mg
  Other Names: Amosartan Tab. 5/50 mg, Amosartan Tab. 5/100 mg
Drug: Amlodipine/Losartan/Chlorthalidone — Amlodipine 5 mg/Losartan Potassium 100 mg/Chlorthalidone 12.5 mg
  Other Names: Amosartan Plus Tab. 5/100/12.5 mg
Drug: current treatment — treatment is done by maintaining the current treatment
  Arms: The usual care group

SUMMARY:
To compare changes in Left Ventricular Mass (LVM) depending on each blood pressure regulation between the intensive care group and the usual care group for patients with hypertension accompanied by aortic valve disease and evaluate an influence of blood pressure regulation on improvement of left ventricular hypertrophy and its safety

DETAILED DESCRIPTION:
1.Primary objectives

- To evaluate changes from baseline in LVM at V5 (24M)

2.Secondary objectives

1. To evaluate changes from baseline in LV global longitudinal strain at V5 (24M)
2. To evaluate changes from baseline in E/E' (E: early diastolic LV inflow velocity, E': early diastolic mitral annulus velocity) at V5 (24M)
3. To evaluate changes from baseline in LV volumes, a stroke volume index and LV ejection fraction at V5 (24M)
4. To evaluate a rate of disease progression

   * In case of Aortic stenosis (AS), to evaluate changes from baseline in Aortic Valve Area (AVA), Vmax, Mean Pressure Gradient (PG) and Valvulo-arterial impedance (Zva) at V5 (24M)
   * In case of Aortic regurgitation (AR), to evaluate changes from baseline in Vena contracta at V5 (24M)
5. To evaluate changes from baseline in blood pressure at V2(6M), V3(12M), V4(18M) and V5(24M)
6. To evaluate a cumulative incidence rate for each visit time point

   * Death, Cardiovascular(CV) death, Heart Failure(HF), Myocardial Infarction(MI), Hospitalization, Aortic Valve Replacement(AVR)
7. To evaluate outcomes of adverse events, physical examination, vital signs (pulse) and laboratory tests (hematological examination, blood biochemical examination, urine test and pregnancy test)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 19 years and < 80 years
2. Diagnosis of mild-moderate AS or mild-moderate AR
3. Applicable to 2.0~3.9 m/s of aortic jet velocity for mild-moderate AS or to 0.2~0.6 cm of Vena contracta for mild-moderate AR
4. Diagnosis of hypertension (SBP > 130 mmHg if being treated or SBP > 140 mmHg if being untreated)
5. For females of childbearing potential; negative pregnancy test results during the screening period and prior to administration of the investigational product, and agreement on use of medically allowable contraceptive measures (condom, oral contraceptive pills, injectable or implantable contraceptives, intrauterine devices, birth control patches, etc.) during the study period
6. Voluntary written consent to taking part in the clinical study and willingness to comply with requirements of the study

Exclusion Criteria:

1. History of a cardiac valve replacement surgery (replacement surgery of mitral valve, aortic valve or tricuspid valve)
2. Accompanied by severe mitral regurgitation
3. Admitted to needing a surgery by the current treatment guidelines
4. Accompanied by symptoms such as angina pectoris, exertional dyspnea, syncope, etc.
5. < 50% of left ventricular ejection fraction
6. History of hypersensitivity reaction to active ingredients of the investigational product (Amlodipine, Losartan and Chlorthalidone), dihydropyridine derivatives, thiazide drugs and other sulfonamide derivatives or their compositions
7. Pregnant or breastfeeding
8. Symptomatic orthostatic hypotension
9. Severe liver failure or renal failure (< 30 mL/min of creatinine clearance)
10. Hereditary angioedema or history of angioedema at treatment with ACE inhibitors or angiotensin II receptor blockers
11. Primary hyperaldosteronism
12. Genetic problems such as galactose intolerance, Lapp Lapp lactase deficiency or glucose-galactose malabsorption
13. Anuria
14. Refractory hypokalemia
15. Hyponatremia or hypercalcemia
16. Symptomatic hyperuricemia (history of gout or uric acid lithiasis)
17. Untreated Addison's disease
18. Appropriately uncontrolled diabetes
19. Congenital or incurable hypertension
20. Diagnosis of severe cerebrovascular disorders (stroke, cerebral infarction, cerebral hemorrhage, etc.) within six months prior to the date of ICF obtainment
21. Wasting disease, autoimmune disease or connective tissue disease
22. Diagnosis of malignant tumor within five years prior to the date of ICF obtainment
23. Administration of another investigational product within four weeks prior to the date of ICF obtainment
24. For a patient who is taking anticoagulants and thrombolytic agents; considered difficult to keep a stable dosage/regimen by the investigator.
25. Considered unsuitable to be a subject by the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
To evaluate changes from baseline in Left Ventricular Mass at 24M | 24 months
  To evaluate changes from baseline in Left Ventricular Mass at 24M

SECONDARY OUTCOMES:
Changes from baseline in Left Ventricular global longitudinal strain at 24M | 24 months
  Changes from baseline in Left Ventricular global longitudinal strain at 24M
Changes from baseline in E/E' (E: early diastolic LV inflow velocity, E': early diastolic mitral annulus velocity) at 24M | 24 months
  Changes from baseline in E/E' (E: early diastolic LV inflow velocity, E': early diastolic mitral annulus velocity) at 24M
Changes from baseline in Left Ventricular volumes at 24M | 24 months
  Changes from baseline in Left Ventricular volumes at 24M
Rate of disease progression | 24 months
  * In case of Aortic Stenosis, to evaluate changes from baseline in Aortic Valve Area, tricuspid regurgitation velocity, Mean Pressure Gradient and Valvulo-arterial impedance at 24M
  * In case of Aortic Regurgitation, to evaluate changes from baseline in Vena contracta at 24M
To evaluate changes from baseline in systolic blood pressure at 6M, 12M, 18M, 24M | 6 months, 12 months, 18 months, 24 months
  To evaluate changes from baseline in systolic blood pressure at 6M, 12M, 18M, 24M
Cumulative incidence rate for each visit time point | 6 months, 12 months, 18 months, 24 months
  Cumulative incidence rate for each visit time point
  - Death, Cardiovascular death, Heart Failure, Myocardial Infarction, Hospitalization, Aortic Valve Replacement
Changes from baseline in stroke volume index at 24M | 24 months
  Changes from baseline in stroke volume index at 24M
Changes from baseline in Left Ventricular ejection fraction at 24M | 24 months
  Changes from baseline in Left Ventricular ejection fraction at 24M

OTHER OUTCOMES:
Occurrence and frequency of adverse events | 6 months, 12 months, 18 months, 24 months
  Occurrence and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, Principal Investigator — 10 institutions including Asan Medical Center
Locations (1):
- 10 Institutions Including Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data

REFERENCES:
- [Derived] Kim M, Choi JH, Kim HK, Kim HL, Shin SH, Jang JY, Park JH, Kim KH, Hong GR, Park SM, Lee SA, Kang DH. Effects of intensive blood pressure control on left ventricular hypertrophy in aortic valve disease. Am Heart J. 2024 Feb;268:45-52. doi: 10.1016/j.ahj.2023.11.012. Epub 2023 Nov 23. PMID 38006908
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623